CLINICAL TRIAL: NCT03780569
Title: A Prospective Trial of NovoTTF-200A Together With Temozolomide and Radiotherapy in Patients With Newly Diagnosed GBM
Brief Title: TTFields Together With Temozolomide and Radiotherapy in Patients With Newly Diagnosed GBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICH-1
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; TTFields; Tumor Treating Fields; Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NovoTTF-200A/Radiotherapy/Temozolomide (Experimental): Patients will receive multiple 1 month courses of continuous NovoTTF-200A treatment together with standard Radiotherapy/Temozolomide followed by maintenance Temozolomide.
  Interventions: Device: NovoTTF-200A; Radiation: Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Device: NovoTTF-200A — Patients receive continuous TTFields treatment using the NovoTTF-200A device. TTFields treatment will consist of wearing four electrically insulated electrode arrays on the scalp. The treatment enables the patient to maintain regular daily routine.
Radiation: Radiotherapy — 60Gy given in 30 2Gy fractions concomitant to temozolomide
Drug: Temozolomide — Temozolomide(TMZ) will be administered at 75 mg/m^2 concomitant to radiotherapy(RT) and NovoTTF-200A.
  Maintenance treatment is to begin about 4 weeks after the end of TMZ/RT/NovoTTF-200A. TMZ is administered at the conventional dosing regimen for 5 days, every 28 days (i.e. 5 days of therapy, 23 days of rest). Cycle 1 is to be given at a dose of 150 mg/m^2 p.o. daily x 5 days, dose to be escalated to 200 mg/m^2 in the absence of toxicity.

SUMMARY:
The study is a prospective, single arm open label study, designed to test the to evaluate the tolerability and safety outcome of newly diagnosed GBM patients treated with NovoTTF-200A concomitant to Radiotherapy/Temozolomide followed by Temozolomide. The device is a portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST CLINICAL EXPERIENCE:

A phase III trial of Optune® (200 kHz) as monotherapy compared to active chemotherapy in recurrent glioblastoma patients showed TTFields to be equivalent to active chemotherapy in extending survival, associated with minimal toxicity, good quality of life, and activity within the brain (14% response rate). In addition, a phase III trial of Optune® combined with maintenance temozolomide compared to maintenance temozolomide alone has shown that combined therapy led to a significant improvement in both progression free survival and overall survival in patients with newly diagnosed glioblastoma without the addition of high grade toxicity and without decline in quality of life.

DESCRIPTION OF THE TRIAL:

All patients included in this trial are newly diagnosed GBM patients who underwent a biopsy or surgery. In addition, all patients must meet all eligibility criteria.

Eligible patients will be enrolled to receive Radiotherapy(RT)/Temozolomide/NovoTTF-200A followed by maintenance TMZ and NovoTTF-200A.

Baseline tests will be performed, The patients will be treated continuously with the device until second progression. They will possibly receive a second line treatment that can be one of the following: re-operation, local radiotherapy (gamma-knife), a second line of chemotherapy or a combination of the above.

NovoTTF-200A treatment will consist of wearing four electrically insulated electrode arrays on the head. Electrode array placement will require shaving of the scalp before and frequently during the treatment. After an initial short visit to the clinic for training and monitoring, patients will be released to continue treatment at home where they can maintain their regular daily routine.

During RT, patients will be seen twice a week and the arrays will be removed to inspect the skin condition. In addition during the trial, patients will need to return once every month to the clinic where an examination by a physician and a routine laboratory examinations will be done. These routine visits will continue for as long as the patient's disease is not progressing for the second time under the study treatment. If such occurs, patients will need to return once per month for two more months to the clinic for similar follow up examinations.

During the visits to the clinic patients will be examined physically and neurologically. Additionally, routine blood tests will be performed. A routine MRI of the head will be performed at baseline and every second month thereafter, until second progression. After this follow up plan, patients will be contacted once per month by telephone to answer basic questions about their health status.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (200 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by Novocure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause electrically-charged cellular components of these cells to change their location within the dividing cell, disrupting their normal function and ultimately leading to cell death. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields interfere with the normal orientation of these tiny motors related to other cellular components since they are electrically-charged as well. As a result of these two effects, tumor cell division is slowed, results in cellular death or reverses after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach. Finally, the frequency of TTFields applied to each type of cancer is specific and may not damage normally dividing cells in healthy tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of GBM according to WHO classification criteria.
2. Supratentorial tumor location
3. Age ≥ 18 years
4. Recovered from maximal debulking surgery, if applicable (gross total resection, partial resection and biopsy-only patients are all acceptable)
5. Planned standard adjuvant chemoradiotherapy of approx. 60 Gy of Radiotherapy (RT), or biologically equivalent dose, according to local practice, and concomitant Temozolomide (TMZ) chemotherapy (75mg/m^2 daily). Any other cytotoxic or biologic anti-tumor therapy received prior to enrollment will be considered an exclusion.
6. Planned treatment with adjuvant/maintenance TMZ (150-200 mg/m^2 daily x 5 d, q28 days)
7. Karnofsky performance status ≥ 70
8. Life expectancy ≥ 3 months
9. Participants of childbearing age must use effective contraception.
10. All patients must sign written informed consent.
11. NovoTTF-200A treatment start date at least 2 weeks out from brain surgery.
12. NovoTTF-200A treatment start prior to or at the beginning of RT/TMZ
13. Stable or decreasing dose of corticosteroids for the last 7 days prior to enrollment, if applicable.

Exclusion Criteria:

1. Participation in another clinical treatment trial
2. Pregnancy or breast feeding
3. Significant co-morbidities at baseline which would preclude TMZ treatment
4. Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
5. Infra-tentorial tumor location
6. Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
7. History of hypersensitivity reaction to TMZ or a history of hypersensitivity to DTIC.
8. Known allergies to medical adhesives or gel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-04-27 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Safety of concomitant Radiotherapy/Temozolomide with NovoTTF-200A: The incidence of Radiotherapy treatment delays during concomitant Radiotherapy/Temozolomide/NovoTTF-200A will be documented including severity and relationship to NovoTTF-200A. | 2 years
  The incidence of Radiotherapy treatment delays during concomitant Radiotherapy/Temozolomide/NovoTTF-200A will be documented including severity and relationship to NovoTTF-200A.

SECONDARY OUTCOMES:
Progression free survival | 2 years
Overall survival | 2 years
Adverse events, severity and frequency | 2 years
  Safety of NovoTTF-200A treatment based on the incidence and severity of adverse events and toxicities.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225